CLINICAL TRIAL: NCT07375797
Title: Fecal Microbiota Transplantation Intervention on Microbiota Composition and Insulin Sensitivity in Diabetes
Acronym: FeMIC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Jutland Regional Hospital (Other)
Collaborators: Steno Diabetes Center Aarhus (SDCA), Aarhus University Hospital (Unknown); Aarhus University Hospital (Other); University of Aarhus (Other)
Responsible Party: Principal Investigator, Henrik Holm Thomsen, Consultant Endocrinologist, Central Jutland Regional Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1-10-72-140-23
Record Dates: First submitted 2026-01-12; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus Type 2; Fecal Microbiota Transplantation (FMT); Oral Glucose Tolerance Test; Continuous Glucose Monitoring
Keywords: Fecal Microbiota Transplantation; FMT; Insulin Sensitivity; Type II Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fecal Microbiota Transplantation (Experimental): The participants will receive two rounds of FMT with two weeks between each treatment.
  Interventions: Other: Fecal Microbial Transplantation
- Placebo (Placebo Comparator): Placebo capsules visually identical to FMT capsules
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Fecal Microbial Transplantation — The capsules consists of approximately 50 grams of donor feces. This is cryopreserved, homogenized and dispensed into double-coated, acid resistant enterocapsules. A single treatment includes approximately 25 capsules.
  The fecal material is obtained from healthy donors, recruited from thoroughly screened healthy blood donors and processed in compliance with the European Tissue and Cells Directive. Further, the donors lipid status and HbA1c is screened, ensuring only metabolically healthy donors are included.
  Other Names: FMT
  Arms: Fecal Microbiota Transplantation
Other: Placebo — The placebo products consists of the same capsules as FMT. The content of the capsules is produced from a suspension of glycerol, saline and food coloring. The number of placebo capsules will correspond to the amount of FMT capsules.
  The placebo capsules will be identical in visual appearance.
  Other Names: Placebo capsules
  Arms: Placebo

SUMMARY:
The purpose of the trial is to investigate the effect of fecal microbiota transplantation versus placebo on glycemic metabolism and gut microbiota composition in people with type 2 diabetes.

DETAILED DESCRIPTION:
People with type 2 diabetes have been shown to exhibit an altered composition of the gut microbiota, including a reduced abundance of butyrate-producing bacteria. Although the underlying mechanisms are not fully elucidated, alterations in gut microbiota composition may be important in the pathogenesis of type 2 diabetes and in metabolic regulation. Fecal microbiota transplantation (FMT) from lean donors has been shown to transiently improve insulin sensitivity and increase the abundance of butyrate-producing bacteria in individuals with metabolic syndrome.

A double-blinded, randomized, placebo-controlled trial will be conducted to investigate the effects of FMT on glycaemic metabolism and gut microbiota composition in individuals with type 2 diabetes. A total of 16 participants will be randomly assigned to one of two groups, receiving either FMT or placebo.

Glycaemic metabolism will be assessed at baseline and again at week 7 post-intervention using three complementary measures: the Homeostatic Model Assessment of Insulin Resistance (HOMA-IR), an oral glucose tolerance test (OGTT) for the Matsuda index, and continuous glucose monitoring (CGM). In addition, stool samples will be collected before and after the intervention to evaluate changes in gut microbiota composition following FMT, for example using 16S rRNA gene sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Has type 2 diabetes

Exclusion Criteria:

* Treatment with insulin or sulfonylurea drugs.
* Treatment with antibiotics, probiotics/lactic acids cultures, or proton pump inhibitors within the last three months.
* Regular exercise and/or more than 150 minutes of moderate intensity exercise or 75 minutes of high intensity exercise per week, within the last 6 months.
* Diagnosed with unstable angina, recent (within the last 8 weeks) myocardial infarction, any disease in the coronal arteries, decompensated heart failure (NYHA II-IV), severe valvular disease, lung disease
* Hypertension which is not currently under medical control (systolic pressure >200 mmHg and/or diastolic pressure >130 mmHg)
* Bariatric surgery within the previous year or a plan to undergo bariatric surgery during the study period
* Self-reported drug or alcohol abuse
* Patients preparing for or currently experiencing pregnancy during the study period
* Disease of the liver and/or gallbladder, including parenchymal liver disease, liver cirrhosis, pancreatitis, autoimmune liver disease
* All diseases of the gastrointestinal tract, which can lead to or increase the risk of defects in the mucosal membrane. This includes chronic diarrhea, inflammatory bowel disease, malabsorption, malnutrition, recent infection with clostridium difficile, primary sclerosing cholangitis, radiation induced enteritis, chemotherapy induced diarrhea, hematological diseases
* Reactive hypoglycemia
* Anemia and other diseases of the bone marrow
* Kidney diseases, including moderate albuminuria and other disturbances in the electrolytes balance
* Food allergies, allergies towards catheters (i.e. Venflon) and other instruments used in the study.
* Other condition deeming individuals inappropriate for recruitment according to the investigators or sponsor

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity | At baseline and at week 7
  Insulin sensitivity assessed by the Matsuda index, calculated from plasma glucose (in mmol/L) and serum insulin(in pmol/L) concentrations measured repeatedly during a standardized oral glucose tolerance test at baseline and after 7 weeks.

SECONDARY OUTCOMES:
Time-in-range | At baseline and at week 7
  Percentage of time with interstitial glucose values between 3.9 and 10.0 mmol/L, derived from continuous glucose monitoring data collected over a 10-day period at baseline and during the final two weeks of the intervention.
Hemoglobin A1c | At baseline and at week 7
  Hemoglobin A1c in plasma (in mmol/mol)
Glucose management indicator | At baseline and at week 7
  Glucose management indicator (GMI) calculated from mean interstitial glucose values derived from continuous glucose monitoring data collected over a 10-day period at baseline and during the final two weeks of the intervention.
Body mass index | At baseline and at week 7
  Weight (in kilograms), height (in meters) for calculation of BMI
Waist circumference | At baseline and at week 7
  Waist circumference(in centimeters)
Microbiome analysis | At baseline and at week 7
  Fecal samples will be collected and analyzed to characterize the gut microbiome and its changes in response to the intervention. Analyses may include 16S rRNA gene sequencing and/or other molecular or biochemical methods to assess microbial composition, diversity, and selected functional features. The specific analytical methods will be defined prior to analysis.

OTHER OUTCOMES:
LEAP-2/ghrelin | At baseline and at week 7
  LEAP-2/ghrelin (arbitrary units, with LEAP-2 and ghrelin in ng/ml)
GLP-1 | At baseline and at week 7
  glukagonlike peptide-1 (in pmol/l)
Interleukin 1-beta | At baseline and at week 7
  IL1B measured with Multiplex (in pg/ml)
Triglycerides | At baseline and at week 7
  Measurements of serum triglycerides (in mmol/L)
C-reactive protein | At baseline and at week 7
  C-reactive protein (mg/L))
Remnant cholesterol | At baseline and at week 7
  Remnant is calculated from Total, LDL, and HDL-cholesterol (all in mmol/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Diagnostics Center, Regional Hospital Central Jutland (HEM), Viborg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared upon reasonable request to the corresponding author. Data will be de-identified where possible and made available to qualified researchers for scientific purposes. Due to the small sample size and risk of re-identification, data will not be deposited in a public repository
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available beginning after publication of the primary study results and will remain available for a reasonable period thereafter, subject to continued data governance and ethical approval.
Access Criteria: Access to IPD and supporting information will be granted to qualified researchers with a scientifically sound research proposal. Requests will be reviewed by the study investigators. Approved users will receive access to de-identified data relevant to the approved analysis, following execution of a data use agreement. Data will be shared via secure data transfer. Due to the small sample size, full datasets will not be made publicly available.

REFERENCES:
- See also: Centre for Faecal Microbiota Transplantation - CEFTA — https://cefta.au.dk/